CLINICAL TRIAL: NCT00448578
Title: A Double Dummy & Double Blind, Multicenter, Randomized Study of the Efficacy and Safety of Seroquel (Quetiapine Fumarate) and Lithium as Monotherapy in the Treatment of Acute Mania in Patients With Bipolar Disorder
Brief Title: Efficacy and Safety of Seroquel and Lithium as Monotherapy in Acute Mania Treatment in Bipolar Disorder Patients
Acronym: STAR
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: D1440L00006
Record Dates: First submitted 2007-03-16; First posted 2007-03-19 (Estimated); Last update posted 2010-12-09 (Estimated); Status verified 2010-12

CONDITIONS: Mania; Bipolar Disorder
Keywords: Acute Mania
MeSH Terms: conditions — Mania; Bipolar Disorder | interventions — Quetiapine Fumarate; Lithium

INTERVENTIONS:
Drug: Quetiapine Fumarate
Drug: Lithium

SUMMARY:
This is a randomised, double blind, double dummy, multicentre, parallel-group study to compare the efficacy and safety of quetiapine and lithium used as monotherapy in the treatment of mania in patients hospitalised for an acute manic episode. After given of informed consent and undergoing screening procedures, the patients will be randomised into quetiapine or lithium group on Day 1. The efficacy of study treatment on symptoms of mania will be assessed at Day 28. Patients will not permitted to use any psychoactive or antipsychotic medications throughout the study period other than those expressly permitted by the protocol. The patients are required to be hospitalised for the treatment and assessment defined in the protocol. He/She could be discharged from the hospital after Week 2 (i.e. On Day 15) if the investigator believes that it will be clinical appropriate to discharge the patient, that the patient is not suicidal or homicidal, and that the patient could reasonably be expected to continue in the study on an outpatient basis. The patients discharged after Day 15 will be given sufficient study medication for the period from discharge to the next visit. At each centre, the same individual will administer a specific psychiatric assessment for a patient at all study visits in order to reduce variability in rating scale scoring. Before the initiation of the study, a consistency assessment will be done among the investigators who conduct the scale assessment in each centre.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent for study participation, signed by the patient's legal guardian.
* Both at screening and at randomization (Day 1), had a YMRS total score of at least 20.

Exclusion Criteria:

* Known intolerance or lack of response to quetiapine or lithium, as judged by the investigator.
* Known or suspected hypersensitivity to quetiapine or lithium.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150
Dates: Start 2005-08; Study Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
Effectiveness of quetiapine fumarate used as monotherapy in treatment of symptoms of acute mania in patients with bipolar disorder by evaluation of the change from baseline in YMRS total score at Day 28 using the last observation carried forward method

SECONDARY OUTCOMES:
The effectiveness of quetiapine used as monotherapy to treat symptoms in patients with acute mania by evaluation of YMRS response rate at Day 28 (LOCF).

CONTACTS AND LOCATIONS:
Overall Officials: Clara Gu, Study Chair — AstraZeneca
Locations (6):
- China (6):
  - Research Sites, Beijing
  - Research Site, Guangzhou
  - Research Site, Kunming
  - Research Site, Nanjing
  - Research Site, Shanghai
  - Research Site, Wuhan